CLINICAL TRIAL: NCT01491386
Title: A Clinical Investigation of Recombinant Human Bone Morphogenetic Protein-2 and Absorbable Collagen Sponge With the LT-CAGE® Device for Anterior Lumbar Interbody Fusion in Patients With Symptomatic Degenerative Disc Disease
Brief Title: Pivotal Study of rhBMP-2/ACS/LT-CAGE® Device for Anterior Lumbar Interbody Fusion in Patients With Symptomatic Degenerative Disc Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-9702
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Degenerative Disc Disease
Keywords: symptomatic degenerative disc disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhBMP-2/ACS (Experimental)
  Interventions: Device: rhBMP-2/ACS/LT-CAGE® Device
- Autogenous Bone (Active Comparator)
  Interventions: Device: Autogenous Bone/LT-CAGE® Device

INTERVENTIONS:
Device: rhBMP-2/ACS/LT-CAGE® Device — LT-CAGE® device with recombinant human bone morphogenetic protein-2 ( rhBMP-2) and the absorbable collagen sponge (ACS).
  Other Names: Recombinant human bone morphogenetic protein
  Arms: rhBMP-2/ACS
Device: Autogenous Bone/LT-CAGE® Device — LT-CAGE® device with autogenous bone taken from the iliac crest.
  Other Names: Autograft
  Arms: Autogenous Bone

SUMMARY:
This study is designed to assess the safety and effectiveness of the rhBMP-2/ACS/LT-CAGE® device as compared to the LT-CAGE® device with autogenous bone in patients with symptomatic degenerative disc disease using an open surgical technique.

ELIGIBILITY:
Inclusion Criteria:

1. Has degenerative disc disease as noted by back pain of discogenic origin, with or without leg pain, with degeneration of the disc confirmed by patient history ( e.g.,pain [leg, back, or symptoms in the sciatic nerve distribution], function deficit and/or neurological deficit) and radiographic studies ( e.g., CT, MRl, X-Ray, etc.) to include one or more of the following:

   * instability (defined as angular motion > 5° and/or translation >= 4mm, based on Flex/Ext radiographs);
   * osteophyte formation;
   * decreased disc height;
   * thickening of ligamentous tissue;
   * disc degeneration or herniation; and/or
   * facet joint degeneration.
2. Has preoperative Oswestry score > 35.
3. Has no greater than Grade 1 spondylolisthesis utilizing Meyerding's Classification (Meyerding HW, 1932.).
4. Has single-level symptomatic degenerative involvement from L4 to S1.
5. Is at least 18 years of age, inclusive, at the time of surgery.
6. Has not responded to non-operative treatment (e.g., bed rest, physical therapy, medications, spinal injections, manipulation, and/or TENS) for a period of at least 6 months.
7. If female of child-bearing potential, who is not pregnant or nursing, and who agrees to use adequate contraception for 16 weeks following surgery.
8. Is willing and able to comply with the study plan and sign the Patient Informed Consent Form.

Exclusion Criteria:

1. Had previous anterior spinal fusion surgical procedure at the involved level.
2. Has posterior spinal instrumentation (which will not be removed) stabilizing the involved level or has had a previous posterior lumbar interbody fusion procedure at the involved level.
3. Has a condition which requires postoperative medications that interfere with fusion, such as steroids.
4. Has been previously diagnosed with osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated.
5. Has presence of active malignancy.
6. Has overt or active bacterial infection, either local or systemic.
7. ls grossly obese, i.e., weight > 40% over ideal for their age and height.
8. Has fever ( temperature > 101° F oral) at the time of surgery.
9. Has a documented titanium alloy allergy or intolerance.
10. Is mentally incompetent. if questionable, obtain psychiatric consult.
11. Has a Waddell Signs of Inorganic Behavior score of 3 or greater.
12. Is a prisoner.
13. Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug usage.
14. Is a tobacco user at the time of surgery.
15. Has received drugs which may interfere with bone metabolism within two weeks prior to the planned date of spinal fusion surgery (e.g., steroids or methotrexate).
16. Has a history of autoimmune disease (Systemic Lupus Erythematosus or Dermatomyositis).
17. Has a history of exposure to injectable collagen implants.
18. Has a history of hypersensitivity to protein pharmaceuticals (monoclonal antibodies or gamma globulins) or collagen.
19. Has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following rhBMP-2/ACS implantation.
20. Has received any previous exposure to any/all BMP's of either human or animal extraction.
21. Has a history of allergy to bovine products or a history of anaphylaxis.
22. Has history of endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, Ehlers- Danlos syndrome, or osteogenesis imperfecta).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 1998-08; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Overall success | 24 months
  A patient will be considered an overall success if all of the following conditions are met:
  1. fusion;
  2. pain/disability (Oswestry) improvement;
  3. maintenance or improvement in neurological status;
  4. no serious adverse event classified as implant associated or implant/surgical procedure associated;
  5. no additional surgical procedure classified as a "failure."

SECONDARY OUTCOMES:
Disc Height Measurement | 24 months
General Health Status (SF-36) | 24 months
Pain Status (Numerical Rating Scale) | 24 months
Patient Satisfaction | 24 months
Patient Global Perceived Effect | 24 months